CLINICAL TRIAL: NCT06005805
Title: A Study To Evaluate the Feasibility of the Decentralized Clinical Trial in South Korea: to Evaluate the Effect of Mastic Gum in Participants With Functional Dyspepsia Symptoms
Brief Title: A Study To Evaluate the Feasibility of the Decentralized Clinical Trial in South Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Sang Yu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCT-102
Record Dates: First submitted 2023-08-06; First posted 2023-08-23 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Mastic Resin; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mastic gum with dietary modification (Experimental): Mastic gum with dietary modification (for 21 days)
  Interventions: Dietary Supplement: Mastic gum; Behavioral: Dietary modification
- Dietary modification (Placebo Comparator): Dietary modification (for 21 days)
  Interventions: Behavioral: Dietary modification

INTERVENTIONS:
Dietary Supplement: Mastic gum — Mastic gum 3g/pack daily for 21 days
  Arms: Mastic gum with dietary modification
Behavioral: Dietary modification — Adhere to the dietary recommendations for Korean dyspepsia patients

SUMMARY:
The goal of this study is to evaluate the feasibility of a decentralized clinical trial in South Korea. The main questions it aims to answer are:

* Does decentralized elements feasible in Korea?
* Does Mastic gum alleviates symptoms and modifies stool microbiome in Korean patients with functional dyspepsia?

DETAILED DESCRIPTION:
The trial aims to evaluate decentralized elements in South Korea, including clinical laboratory testing using local laboratories, medication adherence assessment using wearable devices, analysis of self-kit specimens, delivery and tracking of investigational medication, real-time remote interview of subjects and e-consent acquisition.

Mastic gum is registered with the Ministry of Food and Drug Safety in South Korea as a dietary supplement for gastric health, and the study aims to explore the effect on the gastrointestinal symptoms and composition of the stool microbiome.

ELIGIBILITY:
1) Inclusion Criteria

1. Adults aged 19 to 75 years old at the time of consent.
2. The sum of the intensity and frequency score of the six major symptoms (epigastric pain, early satiety, postprandial fullness, bloating, belching and nausea) of the self-evaluation questionnaire for dyspepsia (SEQ-DYSPEPSIA) is 12 or more.

2) Exclusion Criteria

1. Those with symptoms (dysphagia, severe dysphagia, bleeding, weight loss, anemia, bloody stools) that may suggest a malignant disease of the gastrointestinal tract.
2. Subjects with a diagnosis of eosinophilic esophagitis or a history of eosinophilic esophagitis.
3. Have or have had clinically significant hepatic, renal, neurologic, respiratory, endocrine, hematologic and oncologic, cardiovascular, urinary, or psychiatric disease.
4. Pregnant or lactating women
5. Have or have had a history of clinically significant hypersensitivity to the dietary supplement to be administered.
6. Aspartate aminotransferase or alanine aminotransferase greater than 5 times the upper limit of normal range on screening tests
7. Subjects who are expected to take other medications within the study period that may affect the evaluation of the effectiveness of the study substance (gastrointestinal motility promoters, acid secretagogues, proton pump inhibitors, nonsteroidal anti-inflammatory drugs, anticholinergics, erythromycin, corticosteroids, antidepressants, etc.
8. Those deemed by the investigator to be unsuitable for participation in the clinical trial due to other reasons.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Specimen delivery time | up to 1 months
  Time from collection at the local laboratory to delivery of specimen and reporting of results
Self-kit success rate | up to 1 months
  Fraction of patients who utilized and delivered a self-test kit on the scheduled date
Adverse event management time | up to 1 months
  In the event of an adverse event requiring medical attention, time from report to response

SECONDARY OUTCOMES:
Self-evaluation questionnaire for dyspepsia (SEQ-DYSPEPSIA) score | baseline, immediately after the intervention
  A self-evaluation questionnaire for dyspepsia score comprised 11 symptoms. Each symptom is measured on a 5-point scale for both frequency and intensity. The total score range from 22 to 110 and higher scores mean a worse outcome.
Gut Microbiome Index | baseline, immediately after the intervention
  An index that combines microbial diversity, the proportion of pro-inflammatory microbes, the proportion of microbes that produce anti-inflammatory substances, and similarity to hunter-gatherers.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Huh KY, Chung JY, Yu KS. Methodology for Assessing Patient Centricity and Data Integrity in Clinical Trials With Decentralized Elements: A Pilot Trial on Mastic Gum. Clin Transl Sci. 2025 Sep;18(9):e70343. doi: 10.1111/cts.70343. PMID 40903850